CLINICAL TRIAL: NCT05255419
Title: "OnCall": Implementing a Mobile Health Approach to Post-traumatic Stress Injury (PTSI) Prevention and Peer Support for Canadian Public Safety Personnel
Brief Title: "OnCall": Implementation Study of M-Health for Canadian Public Safety Personnel
Acronym: OnCall
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Collaborators: Movember Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 13990
Record Dates: First submitted 2022-02-16; First posted 2022-02-24 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Mental Health Issue; Mental Stress; Post Traumatic Stress Disorder
Keywords: peer support; mobile health
MeSH Terms: conditions — Stress, Psychological; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: OnCall mobile health peer support app — Mobile health platform that provides anonymous access to peer support services that has been co-design by and for Canadian public safety personnel. OnCall is for frontline public safety providers; features include links to mental health self-assessment tools, a wellness toolbox, "tips to cope" articles and peer wisdom videos, and options to reach out to a peer support provider of their choice via telephone or text. The OnCallSupport app is for the peer support providers which includes a list of resources and an opportunity to create post-action reports following the peer support encounter. Connections are made to peer support via a telephone service that disguises the contact information of both parties. The app platform includes options to complete feedback surveys related to the app and to the peer support encounter.
  Other Names: OnCall, OnCallSupport

SUMMARY:
First Responders, or Public Safety Personnel (PSP), play a key role in protecting the health and safety of Canadians, yet this important work can take a toll on their mental health, leading to an elevated risk of post-traumatic stress injury (PTSI). Mobile health approaches are a promising tool to facilitate access to confidential on-demand mental health support both when and where it is needed. There are gaps, however, in evidence to support the use of m-health apps, particularly in relation to implementation in the PSP community.

The overall purpose of this prospective cohort implementation study is to explore how OnCall, a new mobile health peer-to-peer support application for Public Safety Personnel (PSP) affects peer support help-outreach in the workplace. Implementation and impact will be tracked over 6-month period in a purposive sample of 6-8 different PSP organizations across Canada. Study findings will inform recommendations for optimizing implementation of the m-health platform with employees in other PSP organisations.

DETAILED DESCRIPTION:
Public Safety Personnel (PSP), including, but not limited to correctional workers, emergency communications, firefighters, paramedics, and police officers have an elevated risk of post-traumatic stress injury (PTSI) due to the challenging nature of their work. Unfortunately, they also face barriers to seeking support due to stigma combined with gendered beliefs regarding perception of weakness, pressure to control emotions and reluctance to seek help, as well as lack of access to timely, high-quality care, particularly for those who work in rural or remote areas. Peer support is highly valued, however peer support services are often fragmented with inconsistencies in training and varied models of service delivery, and there are almost no systematic evaluations to inform continuous improvements. Mobile health technology (m-health apps) can be an effective and efficient approach to reaching large numbers of PSP, regardless of location, and an accessible conduit to peer (and professional) support. This research study will explore the implementation and impact of a new m-health platform (OnCall and OnCallSupport) that is customized for public safety personnel.

There are two sets of research questions guiding this project. The first set relates to implementation; How do frontline PSP utilize the OnCall support app? How do these patterns of use change over time? What organizational and social forces shape patterns of app use? The Consolidated Framework for Implementation Research (CFIR) will be used to guide data collection and analysis of the app implementation. The second set of questions relate to impact of the app on service users. Does use of the app increase outreach to peer support? Does peer support provided in the app reduce levels of mental distress? Does use of the app affect mental health literacy, symptoms of anxiety, depression and post-traumatic stress disorder (PTSD), and/or work performance?

Implementation of the app will be studied over a 6 month period with employees in 6-8 PSP organizations. Organizations will be purposively selected to explore differences in size, geographical location, and type of service. All participating organizations must have an established peer support program, with established training and ongoing support for the peer providers. The organizations must also identify 1-2 organizational champions who will liaise with the research team, organizational leaders and frontline employees. Peer providers within the organization will be oriented to the OnCallSupport app, and asked to provide support via this m-health platform. All employees in each organization will then be invited to download the OnCall app via tokens provided by the research team. No personal data is collected in the app, and connections with the peer providers are completely private. Employees will also be invited to complete baseline, 3 month and 6 month follow-up surveys to track changes in help-outreach, mental health literacy, symptoms of anxiety, depression and PTSD, as well as work performance. Employees are able to use the app without participating in the online surveys.

Data collection will include: a) interviews with champions in each organization at the start and end of the 6-month trial, b) surveys with app users at baseline, 3-month and 6-months, c) review of anonymous, aggregate app utilization data, over the trial period and d) focus group discussions with peer support providers at 1 month and 6 months.

Analysis of the implementation data (interview transcripts with organizational champions, focus group transcripts with peer support providers, and software analytics re: patterns of app use) will be informed by the CFIR framework to identify how the outer setting, inner setting, the intervention, participants and process of implementation affect how employees respond to the app.

Analysis of the impact data will include evaluation of whether there is a significant change over time in each of the outcomes (help-outreach, mental health literacy, symptoms of anxiety, depression, PTSD, work performance). Pre/post data from the baseline, 3- and 6-month follow-up surveys will be compared to track changes in dimensions of mental health literacy, levels of mental distress(standardized assessments of anxiety, depression, PTSD), and frequency of outreach behaviors in seeking mental health support. Data will be compared across organizations to highlight links between implementation and outcomes. Multiple hierarchical linear regression analyses will be conducted to examine differences in effectiveness based on gender, service, job tenure. Demographic variables will be used as primary step independent variables, with each primary outcome variable set as the dependent variable for a dedicated regression. The investigators will include a sex and gender-based analysis (SGBA) since biological sex and socially constructed gender can affect stress responses, mental health, and help outreach. Gender is particularly important with respect to peer support needs, engagement with technology, and mental health outcomes. In keeping with Sex and Gender Equity in Research (SAGER) guidelines, gender will be considered throughout the design and analysis. In both quantitative and qualitative analyses, gender will be considered as a potential mediator. For regression modelling, gender will be included as a covariate, considering interactions between gender and other variables, and where possible disaggregated modelling will be conducted for men and women to determine if differences exist.

Analysis from all data sources will be used to generate recommendations for optimizing implementation and impact at an individual and organization level.

ELIGIBILITY:
Inclusion Criteria:

* Public Safety providers (police, fire, paramedics, corrections, emergency communications)
* Employed (full or part-time) by the participating organizations
* Agree to download the OnCall app on their mobile phone (Android or Apple)

Exclusion Criteria:

* Not able to access app on their mobile health device

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals employed by participating Public Safety Organizations (corrections, EMS, police, emergency communications, fire)
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2022-07-30 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Accessing peer support via phone or text via the OnCall app (frequency count) | Monthly intervals from 1 to 6 months
  Number of times OnCall users initiates a text or phone call to peer support service via the app platform (software analytics)

SECONDARY OUTCOMES:
Change in Mental health literacy (7-point Likert scale rating) | baseline, 3 months, 6 months
  Rating using a 7 point Likert scale of perceived improvement in knowledge of how to identify and address mental health issues. Range 0-7 with higher scores indicating higher levels of perceived literacy.
Change in level of distress (Visual analogue scale) | Immediately following a peer support call or text exchange via the app
  Following peer support encounter, a pop-up survey in the app asks users to rate their level of distress before and after the encounter using a 100-point Visual Analogue scale
Changes in symptoms of anxiety (GAD-2 screening tool) | baseline, 3 months, 6 months
  The Generalised Anxiety Disorder (GAD-2) scale is a 2-item screening tool for anxiety; scores range from 0-6 with a score of 3 or more as indicative of potential generalized anxiety disorder
Change in symptoms of depression (PHQ-2 screening tool) | baseline, 3 months, 6 months
  The Patient Health Questionnaire (PHQ-2) is a 2-item screening tool for depression; score ranges from 0-6, with a score of 3 or more as indicative of major depression.
Change in symptoms of trauma (PTSD Checklist - PCL-5) | baseline, 3 months, 6 months
  The Post-Traumatic Stress Disorder Checklist (PCL-5) is a 20-item self-report measure that assesses the presence and severity of PTSD symptoms over the past month. Scores range from 0-80 with higher scores indicating more severe impairment (cut-off scores 31-33).
Change in functioning at work (Lam Employment Absence and Productivity Scale -LEAPS) | baseline, 3 months, 6 months
  The LEAPS is a 10-item, self-rated scale that provides a measure of functioning at work. Scores range from 0-28 with higher scores indicating more significant impairment.
Satisfaction with app (via adapted Mobile Application Rating Scale) | 3 months, 6 months
  The adapted Mobile Application Rating Scale (MARS) asks users to rate app using a 5-point LIkert scale on the following 5 dimensions: engagement, functionality, aesthetics, and information quality; and overall subjective quality. Higher scores indicate greater levels of satisfaction (some reverse scoring)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra E Moll, PhD, Principal Investigator — McMaster University

IPD SHARING:
Plan to Share IPD: Undecided
May share aggregate utilisation data without personal identifiers.